CLINICAL TRIAL: NCT02411916
Title: Effect of Adjunctive Misoprostol on Blood Loss at Vaginal Delivery
Brief Title: Effect of Adjunctive Misoprostol Treatment on Blood Loss at Vaginal Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York City Health and Hospitals Corporation (Other)
Responsible Party: Principal Investigator, Aleksandr Fuks, Directore, Department OB / GYN , Queens Hospital Center, New York City Health and Hospitals Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QHC11-237
Record Dates: First submitted 2015-04-03; First posted 2015-04-08 (Estimated); Results first posted 2021-09-30 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention cases (Experimental): patient receiving misoprostol
  Interventions: Biological: misoprostol
- controls (No Intervention): patients not receiving misoprostol

INTERVENTIONS:
Biological: misoprostol — rectal insertion
  Other Names: cytotec
  Arms: intervention cases

SUMMARY:
This document defines the Clinical Investigation Protocol for a study designed to determine whether blood loss after spontaneous vaginal delivery is altered by the addition of misoprostol administration to the standard use of intravenous oxytocin after delivery. The protocol is an open-label randomized prospective trial to be carried out at Queens Hospital Center.

Blood loss will be measured indirectly by comparing the maternal hemoglobin and hematocrit levels on admission in labor to those obtained within 24 hours after delivery.

DETAILED DESCRIPTION:
Some maternal blood loss normally occurs at the time of vaginal delivery. The best estimates indicate that a loss of approximately 500 mL is average, with a range of about 250-700 mL.[1,2] Some of this bleeding arises from birth canal lacerations or surgical incisions (i.e., episiotomy), but most derives from the vessels exposed in the uterine wall at the placental site once the placenta has separated.

Under normal circumstances, shortly after placental separation intense myometrial contractions occur. These raise the pressure within the myometrial wall above that of the blood pressure in the vessels that traverse it, vessels that opened into the intervillous space. Flow in these vessels is thus mechanically attenuated by myometrial contraction, allowing for the formation of intravascular thrombi.

This mechanism for controlling postpartum uterine blood loss works well most of the time. If, however, the uterus remains hypotonic or atonic after delivery, excessive blood loss can occur. In the worst cases, severe uterine hemorrhage ensues. Postpartum hemorrhage is, in fact, the leading cause of maternal mortality in the world, accounting for at least 100,000 deaths annually.[3] Even in the absence of frank hemorrhage, postpartum blood loss can result in maternal anemia. Recuperation of iron stores to recover from this blood loss takes time, and may not occur, especially in low socioeconomic areas where dietary iron consumption is often deficient, and pregnancies tend to occur in close succession.

Postpartum anemia is a significant contributor to short- and long-term morbidity.[5-7] It increases the risk of infection and poor wound healing. Also, the associated fatigue may interfere with the mother's ability to administer child care and to bond appropriately with her infant. Anemic mothers tend to have more difficulty with nursing, and may produce iron-deficient milk. There is thus a strong rationale to minimize postpartum blood loss.

In most US hospitals, parturients receive a high dose of intravenous or intramuscular oxytocin immediately after delivery. This approach has been shown in several studies to reduce the risk of postpartum hemorrhage, [8-11] and is practiced routinely at Queens Hospital Center. Investigators will employ an intravenous infusion of oxytocin (Pitocin®) at a rate of about 50-100 mU/minute. Despite this approach, there is still substantial blood loss at delivery, based on the investigator's preliminary observations shown below. This provides the rationale to determine whether use of an adjunctive drug, namely misoprostol 600 µg rectally, administered after delivery, might reduce blood loss further than does oxytocin alone, thus decreasing the risk of morbidity related to postpartum anemia.

Preliminary Data The investigators examined the hemograms of a randomly chosen consecutive sample of 53 spontaneous vaginal deliveries performed at Queens Hospital Center .

Among these patients, the admission hemoglobin concentration was 11.9±1.2 g/dL and that on the first postparutum day was 10.9±1.3. The mean fall was 1.02 (95% CI 0.74, 1.29), a statistically significant decrease (P<0.0001). Hematocrit levels fell in parallel, by an average of 7.8% of the predelivery value. The mean fall in hemoglobin and hematocrit levels after delivery (1.02 g/dL and 2.81%) is consistent with an average blood loss of about 500 mL. The consistency of these changes and the small associated variance indicate that the change in hemoglobin and hematocrit levels is a meaningful proxy for the assessment of blood lost during vaginal delivery.

Sample size and analysis

Of the expected 800 subjects in this two-treatment parallel design study, the probability is 90% that the study will detect a treatment difference at a two-sided 0.05 significance level if the difference in hemoglobin concentration between treatments is 0.3 g/dL. This analysis assumes that the standard deviation of the postpartum and intrapartum hemoglobin concentrations is not larger than 1.3 g/dL.

Comparison of intrapartum and postpartum hemoglobin and hematocrit levels will be done using a paired t-test. A probability level of 0.05 will be used as the threshold for significance.

Inclusion and exclusion criteria This study will include adult pregnant women regardless of age. Pregnant minors under the age of 18 will not be eligible.

Patients who meet the inclusion criteria for the study will be identified during their prenatal clinical visits, in early latent-labor, or prior to induction of labor or active labor. Informed consent will be obtained by one of the investigators. Consent will be obtained prior to active labor. The informed consenting process will not be initiated among patients in active labor. It will be determined by the investigator whether the patient will receive oxytocin alone or oxytocin and misoprostol. Both drugs are on formulary and will be available on the Labor and Delivery Unit for immediate use.

Randomization A computer-generated table of random numbers will be used to assign the recruited subject to a group. The patient will be assigned to the intervention group and will receive oxytocin and misoprostol or the patient will be assigned to "oxytocin only" group.

Characteristics of Medication Nature of misoprostol Misoprostol is a synthetic prostaglandin E1 analog. It is marketed primarily as a drug to prevent the development of gastric ulcers associated with use of nonsteroidal anti-inflammatory drugs, and is part of the Queens Hospital Center formulary. Originally marketed as Cytotec®, misoprostol is available in a generic form as tablets containing contain either 100 µg or 200 µg. Misoprostol protects the gastric mucosa through several mechanisms. It also has the property of stimulating myometrial smooth muscle contraction.[12] That effect has resulted in the drug's common use in obstetrics for termination of pregnancy, cervical ripening prior to induction of labor and, in large doses, for prevention and treatment of postpartum hemorrhage from uterine atony. [13-19]

Misoprostol can be administered by oral, sublingual, vaginal or rectal routes. It is well absorbed with all these modes of administration, but detailed pharmacokinetic data exist primarily concerning its oral administration. It is rapidly absorbed, and undergoes prompt de-esterification to its free acid, which is responsible for its clinical activity. Peak plasma levels after oral administration occur after 10-15 min. The half-life is 20-40 minutes. The alpha side chain undergoes beta oxidation and the beta side chain undergoes omega oxidation followed by reduction of the ketone to give prostaglandin F analogs. Excretion is primarily in the urine.

Very little misoprostol appears in breast milk. [20,21] After a single 600 µg oral dose of misoprostol to nursing mothers, misoprostol acid was excreted in breast milk. One hour after dosing, the milk concentration was about 67% of the maternal serum level; by five hours, the misoprostol concentrations in breast milk declined to < 1 pg/mL. While no specific data exist for misoprostol concentrations in colostrum, given the very small ingested volume over the first few hours of life, neonatal exposure to the drug in the investigator's study can be expected to be minimal. There are no published reports of adverse effects of misoprostol in breast-feeding infants of mothers taking misoprostol

Misoprostol is classified by the FDA as a Pregnancy Category X drug. This label is related to its possible association with congenital anomalies when used in the first trimester, as well as its abortifacient properties. In the investigator's study, patients will no longer be pregnant when the participant receives the drug.

It is unknown whether Misoprostol and/or Oytocin are excreted in human milk. There is an unconfirmed relation with Misoprostol and/or Oytocin causing digestive problems, such as diarrhea, and abdominal cramps in breast-fed newborns. Pariticipants will be advised to discard breast mild for the first 24 hours to possibly avoid occurrence.

Study Procedure: All subjects will receive the standard dose of intravenous oxytocin, begun within one minute of delivery. Subjects in the study group who have not incurred any of the post-hoc exclusion criteria (episiotomy, major laceration, etc) will receive a dose of 600 µg of misoprostol in addition to their oxytocin. This will be administered in the form of six 100 µg tablets inserted approximately 2 cm into the anorectal canal by the obstetrician or midwife who has performed the delivery. The common method for administering Misoprostol for postpartum hemorrhaging is rectally for local absorption. Since this study is directed toward prevention instead of treatment, the dosage of 600mg is a lower dosage from the 1000mg administered, as standard practices, for treating postpartum hemorrhaging of more than 500cc estimated blood loss. The patient's vital signs will be recorded after delivery according to standard protocols of the obstetric service. The Data Collection forms will be filled out after the delivery by one of the investigators. The measurement of postpartum hemoglobin and hematocrit (H & H) is automatically ordered at 06:00am for all patients who have delivered the day prior, constituting this measurement at "Postpartum Day 1", which is at a minimum of 6 hours after delivery and is enough time for H & H levels to stabilize.

Within 36 hours of delivery, additional information will be collected from the patient's record, including the postpartum hemogram and information about any symptoms or signs related to the misoprostol.

Misoprostol is classified by the FDA as a Pregnancy Category X drug. This label is related to its possible association with congenital anomalies when used in the first trimester, as well as its abortifacient properties. In the investigator's study, patients will no longer be pregnant when the participant receives the drug.

Data Collection elements:

Age, Ethnicity/Race, Gestational age (in weeks), Number of previous deliveries, Number of Fetus, Body-Mass Index (BMI), Amniotic Fluid Index (AFI), Cephalic presentation, Fetal Heart Rate (FHR), Reported fetal Anomaly, Preeclampsia, Trial of Labor after Cesarean (TOLAC) After Delivery, Caesarean section (during delivery), Epidural, Oxytocin in labor (if yes, number of hours before delivery, Other medication used in labor, Episiotomy, Duration of stage 1, 2, and 3, Degree and place of laceration, Estimated Blood Loss (EBL), Transfusion, Placental Abruption, Birth weight Results - includes Follow-up Data, Hemoglobin and Hematocrit (H& H) on admission and on post- partum day #1, Reported Side effect by patient, Post partum temperature, Reports of shivering, Diagnosis of chorioamnionitis.

Post- partum day #1- data collection Postpartum Day 1 is delineated as the first 12:01am clock time from the time of delivery. Post-partum measurements, such as postpartum hemoglobin and hematocrit (H & H), are taken automatically at 06:00am for all deliveries that occurred before midnight (at least 6 hours prior).

ELIGIBILITY:
Inclusion criteria (A patient will be considered for inclusion in the study if she meets all of the following criteria):

* She has a term (≥37 completed weeks) live singleton gestation in cephalic presentation and has been admitted to the Labor and Delivery Unit
* She is in the latent phase of labor or has been admitted for induction of labor or at prenatal clinic visit
* She has had fewer than four prior vaginal deliveries.
* She reports no allergy to misoprostol.

The following factors or conditions will exclude a patient from consideration as a subject:

* The fetus has a known major fetal malformation or chromosome abnormality
* The gestation is multiple.
* There is a breech or other malpresentation
* The patient reports involvement in another clinical trial currently or previously in this pregnancy.
* The patient is expected to have a cesarean delivery.
* The patient had a prior cesarean delivery.
* There has been an intrauterine fetal death.
* There is polyhydramnios (amniotic fluid index >22 cm).
* Presence of acute or chronic renal disease
* Presence of preeclampsia

Exclusion criteria (Of subjects who enter the study, the development of certain conditions will exclude them post hoc from receiving misoprostol under the protocol, and from the data analysis. These conditions include):

* Unanticipated cesarean delivery.
* Performance of episiotomy (third and fourth degree extensions will be excluded).
* Vaginal or cervical laceration, or perineal laceration of more than second degree in depth.
* Severe postpartum hemorrhage requiring intervention immediately after delivery.
* Uterine rupture
* Placental abruption.
* Patient withdrawal of consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Recruiting only pregnant women prior to child-birth delivery.
Enrollment: 143 (Actual)
Dates: Start 2012-03-30 (Actual); Primary Completion 2019-02-16 (Actual); Study Completion 2019-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandr Fuks, MD, Principal Investigator — Queens Hopsital Center
Locations (1):
- Queens Hospital Center, Jamaica, New York, United States

REFERENCES:
- [Background] Pritchard JA, Baldwin RM, Dickey JC, et al. Blood volume changes in pregnancy and the puerperium, 2. Red blood cell loss and changes in apparent blood volume during and following vaginal delivery, cesarean section, and cesarean section plus total hysterectomy. Am J Obstet Gynecol 1962;84:1271-1282.
- [Background] Sosa CG, Althabe F, Belizan JM, Buekens P. Risk factors for postpartum hemorrhage in vaginal deliveries in a Latin-American population. Obstet Gynecol. 2009 Jun;113(6):1313-1319. doi: 10.1097/AOG.0b013e3181a66b05. PMID 19461428
- [Background] Cohen WR. Hemorrhagic shock in obstetrics. J Perinat Med. 2006;34(4):263-71. doi: 10.1515/JPM.2006.051. PMID 16856813
- [Background] Pontieri-Lewis V. The role of nutrition in wound healing. Medsurg Nurs. 1997 Aug;6(4):187-90, 221; quiz 191-2. PMID 9313545
- [Background] van Ramshorst GH, Nieuwenhuizen J, Hop WC, Arends P, Boom J, Jeekel J, Lange JF. Abdominal wound dehiscence in adults: development and validation of a risk model. World J Surg. 2010 Jan;34(1):20-7. doi: 10.1007/s00268-009-0277-y. PMID 19898894
- [Background] Ezechi OC, Edet A, Akinlade H, Gab-Okafor CV, Herbertson E. Incidence and risk factors for caesarean wound infection in Lagos Nigeria. BMC Res Notes. 2009 Sep 22;2:186. doi: 10.1186/1756-0500-2-186. PMID 19772612
- [Background] Teixeira Mde L, Lira PI, Coutinho SB, Eickmann SH, Lima MC. Influence of breastfeeding type and maternal anemia on hemoglobin concentration in 6-month-old infants. J Pediatr (Rio J). 2010 Jan-Feb;86(1):65-72. doi: 10.2223/JPED.1959. PMID 20151087
- [Background] Chelmow D. Postpartum haemorrhage: prevention. BMJ Clin Evid. 2011 Apr 4;2011:1410. PMID 21463537
- [Background] Elati A, Elmahaishi MS, Elmahaishi MO, Elsraiti OA, Weeks AD. The effect of misoprostol on postpartum contractions: a randomised comparison of three sublingual doses. BJOG. 2011 Mar;118(4):466-73. doi: 10.1111/j.1471-0528.2010.02821.x. Epub 2010 Dec 24. PMID 21199290
- [Background] Soltani H, Hutchon DR, Poulose TA. Timing of prophylactic uterotonics for the third stage of labour after vaginal birth. Cochrane Database Syst Rev. 2010 Aug 4;(8):CD006173. doi: 10.1002/14651858.CD006173.pub2. PMID 20687079
- [Background] Elbourne DR, Prendiville WJ, Carroli G, Wood J, McDonald S. Prophylactic use of oxytocin in the third stage of labour. Cochrane Database Syst Rev. 2001;(4):CD001808. doi: 10.1002/14651858.CD001808. PMID 11687123
- [Background] Gemzell-Danielsson K, Bygdeman M, Aronsson A. Studies on uterine contractility following mifepristone and various routes of misoprostol. Contraception. 2006 Jul;74(1):31-5. doi: 10.1016/j.contraception.2006.03.009. Epub 2006 Apr 27. PMID 16781257
- [Background] Cabrera Y, Fernandez-Guisasola J, Lobo P, Gamir S, Alvarez J. Comparison of sublingual versus vaginal misoprostol for second-trimester pregnancy termination: a meta-analysis. Aust N Z J Obstet Gynaecol. 2011 Apr;51(2):158-65. doi: 10.1111/j.1479-828X.2010.01264.x. Epub 2011 Jan 6. PMID 21466519
- [Background] Enakpene CA, Morhason-Bello IO, Enakpene EO, Arowojolu AO, Omigbodun AO. Oral misoprostol for the prevention of primary post-partum hemorrhage during third stage of labor. J Obstet Gynaecol Res. 2007 Dec;33(6):810-7. doi: 10.1111/j.1447-0756.2007.00661.x. PMID 18001447
- [Background] Nasr A, Shahin AY, Elsamman AM, Zakherah MS, Shaaban OM. Rectal misoprostol versus intravenous oxytocin for prevention of postpartum hemorrhage. Int J Gynaecol Obstet. 2009 Jun;105(3):244-7. doi: 10.1016/j.ijgo.2009.01.018. Epub 2009 Feb 26. PMID 19249048
- [Background] Mansouri HA, Alsahly N. Rectal versus oral misoprostol for active management of third stage of labor: a randomized controlled trial. Arch Gynecol Obstet. 2011 May;283(5):935-9. doi: 10.1007/s00404-010-1466-5. Epub 2010 Apr 27. PMID 20422423
- [Background] Baruah M, Cohn GM. Efficacy of rectal misoprostol as second-line therapy for the treatment of primary postpartum hemorrhage. J Reprod Med. 2008 Mar;53(3):203-6. PMID 18441726
- [Background] Lokugamage AU, Sullivan KR, Niculescu I, Tigere P, Onyangunga F, El Refaey H, Moodley J, Rodeck CH. A randomized study comparing rectally administered misoprostol versus Syntometrine combined with an oxytocin infusion for the cessation of primary post partum hemorrhage. Acta Obstet Gynecol Scand. 2001 Sep;80(9):835-9. doi: 10.1034/j.1600-0412.2001.080009835.x. PMID 11531635
- [Background] Haque N, Bilkis L, Haque N, Bari MS, Haque S. Comparative study between rectally administered misoprostol as a prophylaxis versus conventional intramuscular oxytocin in post partum hemorrhage. Mymensingh Med J. 2009 Jan;18(1 Suppl):S40-44. PMID 19377430
- [Background] Vogel D, Burkhardt T, Rentsch K, Schweer H, Watzer B, Zimmermann R, Von Mandach U. Misoprostol versus methylergometrine: pharmacokinetics in human milk. Am J Obstet Gynecol. 2004 Dec;191(6):2168-73. doi: 10.1016/j.ajog.2004.05.008. PMID 15592308
- [Background] Tang OS, Schweer H, Lee SW, Ho PC. Pharmacokinetics of repeated doses of misoprostol. Hum Reprod. 2009 Aug;24(8):1862-9. doi: 10.1093/humrep/dep108. Epub 2009 Apr 23. PMID 19395364
- [Background] Garris RE, Kirkwood CF. Misoprostol: a prostaglandin E1 analogue. Clin Pharm. 1989 Sep;8(9):627-44. PMID 2507215

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patient declined to participate in study
Period: Overall Study
Arm/Group | Intervention Cases | Controls
Started | 73 | 70
Completed | 73 | 70
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Number of enrolled subjects randomized into the 2 groups. Are presented pregnant women who meet the inclusion criteria.
Groups:
- Intervention Cases: patient receiving misoprostol (rectal insertion)
- Total: Total of all reporting groups
Arm/Group | Intervention Cases | Controls | Total
Number analyzed (Participants) | 73 | 70 | 143
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 73 | 70 | 143
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24 (6) | 25 (6) | 24.5 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 70 | 143
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 73 | 70 | 143
consented and randomized pregnant patients [Count of Participants; unit: Participants] — Presented pregnant patients that were consented and randomized into the 2 groups.
  Participants | 73 | 70 | 143

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin
Time Frame: 1 day after delivery
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Intervention Cases | Controls
Number analyzed (Participants) | 73 | 70
mg/dl | 1.08 (0.484) | 1.20 (0.491)

ADVERSE EVENTS:
Time Frame: 3 years, 3 months
Arm/Group | Intervention Cases | Controls
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/70
Other Adverse Events (participants affected / at risk) | 0/73 | 0/70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-01): https://cdn.clinicaltrials.gov/large-docs/16/NCT02411916/Prot_SAP_000.pdf